CLINICAL TRIAL: NCT00330759
Title: A Randomized, Double-Blind, Multicenter Study of Denosumab Compared With Zoledronic Acid (Zometa) in the Treatment of Bone Metastases in Subjects With Advanced Cancer (Excluding Breast and Prostate Cancer) or Multiple Myeloma.
Brief Title: Study of Denosumab vs. Zoledronic Acid to Treat Bone Metastases in Subjects With Advanced Cancer or Multiple Myeloma.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 20050244
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Results first posted 2014-04-09 (Estimated); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Bone Metastases
Keywords: Bone metastases; lytic bone lesions; advanced cancer; multiple myeloma; lymphoma; solid tumors; skeletal related events; skeletal fractures; spinal cord compressions, radiation to bone; surgery to bone, bisphosphonates; denosumab
MeSH Terms: conditions — Multiple Myeloma; Lymphoma; Spinal Cord Compression | interventions — Denosumab; Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- zoledronic acid (Active Comparator): denosumab placebo with active zoledronic acid
  Interventions: Drug: Zoledronic Acid
- denosumab (Experimental): active denosumab with zoledronic acid placebo
  Interventions: Biological: Denosumab

INTERVENTIONS:
Biological: Denosumab — 120 milligrams by subcutaneous injection every 4 weeks
  Arms: denosumab
Drug: Zoledronic Acid — 4 milligrams intravenous Zoledronic Acid over minimum 15 minutes every 4 weeks
  Other Names: Zometa
  Arms: zoledronic acid

SUMMARY:
The purpose of this study is to determine if denosumab is non-inferior to zoledronic acid (Zometa®) in the treatment of bone metastases (lytic bone lesions from multiple myeloma) in subjects with advanced cancer and multiple myeloma (excluding breast and prostate cancer)

ELIGIBILITY:
Inclusion Criteria:

* Adults with histologically/cystologically confirmed advanced cancers including solid tumors, multiple myeloma, and lymphoma
* Radiographic evidence of at least one bone metastasis (or lytic bone lesion from multiple myeloma); ECOG performance status 0, 1, or 2
* Adequate organ function

Exclusion Criteria:

* Diagnosis of breast or prostate cancer
* Current or prior intravenous bisphosphonate administration
* Current or prior oral bisphosphonates for bone metastases, life expectancy of less than 6 months
* Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1779 (Actual)
Dates: Start 2006-06-01 (Actual); Primary Completion 2009-04-01 (Actual); Study Completion 2011-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Henry D, Vadhan-Raj S, Hirsh V, von Moos R, Hungria V, Costa L, Woll PJ, Scagliotti G, Smith G, Feng A, Jun S, Dansey R, Yeh H. Delaying skeletal-related events in a randomized phase 3 study of denosumab versus zoledronic acid in patients with advanced cancer: an analysis of data from patients with solid tumors. Support Care Cancer. 2014 Mar;22(3):679-87. doi: 10.1007/s00520-013-2022-1. Epub 2013 Oct 26. PMID 24162260
- [Background] Henry DH, Costa L, Goldwasser F, Hirsh V, Hungria V, Prausova J, Scagliotti GV, Sleeboom H, Spencer A, Vadhan-Raj S, von Moos R, Willenbacher W, Woll PJ, Wang J, Jiang Q, Jun S, Dansey R, Yeh H. Randomized, double-blind study of denosumab versus zoledronic acid in the treatment of bone metastases in patients with advanced cancer (excluding breast and prostate cancer) or multiple myeloma. J Clin Oncol. 2011 Mar 20;29(9):1125-32. doi: 10.1200/JCO.2010.31.3304. Epub 2011 Feb 22. PMID 21343556
- [Background] Scagliotti GV, Hirsh V, Siena S, Henry DH, Woll PJ, Manegold C, Solal-Celigny P, Rodriguez G, Krzakowski M, Mehta ND, Lipton L, Garcia-Saenz JA, Pereira JR, Prabhash K, Ciuleanu TE, Kanarev V, Wang H, Balakumaran A, Jacobs I. Overall survival improvement in patients with lung cancer and bone metastases treated with denosumab versus zoledronic acid: subgroup analysis from a randomized phase 3 study. J Thorac Oncol. 2012 Dec;7(12):1823-1829. doi: 10.1097/JTO.0b013e31826aec2b. PMID 23154554
- [Background] Vadhan-Raj S, von Moos R, Fallowfield LJ, Patrick DL, Goldwasser F, Cleeland CS, Henry DH, Novello S, Hungria V, Qian Y, Feng A, Yeh H, Chung K. Clinical benefit in patients with metastatic bone disease: results of a phase 3 study of denosumab versus zoledronic acid. Ann Oncol. 2012 Dec;23(12):3045-3051. doi: 10.1093/annonc/mds175. Epub 2012 Jul 31. PMID 22851406
- [Derived] Abdel-Rahman O. Predictors of skeletal-related events among cancer patients with bone metastases treated with zoledronic acid: a secondary analysis of a randomized study. Expert Opin Drug Saf. 2018 Aug;17(8):757-761. doi: 10.1080/14740338.2018.1497157. Epub 2018 Jul 11. PMID 29972647
- [Derived] Body JJ, Bone HG, de Boer RH, Stopeck A, Van Poznak C, Damiao R, Fizazi K, Henry DH, Ibrahim T, Lipton A, Saad F, Shore N, Takano T, Shaywitz AJ, Wang H, Bracco OL, Braun A, Kostenuik PJ. Hypocalcaemia in patients with metastatic bone disease treated with denosumab. Eur J Cancer. 2015 Sep;51(13):1812-21. doi: 10.1016/j.ejca.2015.05.016. Epub 2015 Jun 17. PMID 26093811
- [Derived] Diel IJ, Body JJ, Stopeck AT, Vadhan-Raj S, Spencer A, Steger G, von Moos R, Goldwasser F, Feng A, Braun A. The role of denosumab in the prevention of hypercalcaemia of malignancy in cancer patients with metastatic bone disease. Eur J Cancer. 2015 Jul;51(11):1467-75. doi: 10.1016/j.ejca.2015.04.017. Epub 2015 May 11. PMID 25976743
- [Derived] von Moos R, Body JJ, Egerdie B, Stopeck A, Brown JE, Damyanov D, Fallowfield LJ, Marx G, Cleeland CS, Patrick DL, Palazzo FG, Qian Y, Braun A, Chung K. Pain and health-related quality of life in patients with advanced solid tumours and bone metastases: integrated results from three randomized, double-blind studies of denosumab and zoledronic acid. Support Care Cancer. 2013 Dec;21(12):3497-507. doi: 10.1007/s00520-013-1932-2. Epub 2013 Aug 22. PMID 23975226
- [Derived] Lipton A, Fizazi K, Stopeck AT, Henry DH, Brown JE, Yardley DA, Richardson GE, Siena S, Maroto P, Clemens M, Bilynskyy B, Charu V, Beuzeboc P, Rader M, Viniegra M, Saad F, Ke C, Braun A, Jun S. Superiority of denosumab to zoledronic acid for prevention of skeletal-related events: a combined analysis of 3 pivotal, randomised, phase 3 trials. Eur J Cancer. 2012 Nov;48(16):3082-92. doi: 10.1016/j.ejca.2012.08.002. Epub 2012 Sep 10. PMID 22975218
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 21 June 2006 through 16 May 2008
Pre-assignment Details: A total of 1779 participants were enrolled in the study. Three participants from one site were excluded from all analyses because Institutional Review Board (IRB) review activities and oversight were not ensured.
Groups:
- Zoledronic Acid: Zoledronic acid 4 mg by intravenous injection with a subcutaneous denosumab placebo once every 4 weeks
- Denosumab: Denosumab 120 mg by subcutaneous injection with an intravenous zoledronic acid placebo once every 4 weeks
Period: Overall Study
Arm/Group | Zoledronic Acid | Denosumab
Started | 890 | 886
Received Investigational Product | 878 | 878
Completed | 178 | 180
Not Completed | 712 | 706
Not completed — Death | 316 | 310
Not completed — Disease progression | 104 | 126
Not completed — Withdrawal by Subject | 143 | 124
Not completed — Adverse Event | 48 | 36
Not completed — Participant request | 31 | 22
Not completed — Lost to Follow-up | 16 | 22
Not completed — Noncompliance | 15 | 17
Not completed — Physician Decision | 1 | 2
Not completed — Protocol deviation | 0 | 2
Not completed — Ineligibility determined | 2 | 1
Not completed — Other | 36 | 44

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Zoledronic Acid | Denosumab | Total
Number analyzed (Participants) | 890 | 886 | 1776
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.6 (10.7) | 59.3 (11.4) | 59.9 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 338 | 298 | 636
  Male | 552 | 588 | 1140
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 770 | 770 | 1540
  Black or African American | 29 | 20 | 49
  Hispanic or Latino | 36 | 49 | 85
  Asian | 44 | 36 | 80
  Japanese | 1 | 3 | 4
  American Indian or Alaska Native | 2 | 0 | 2
  Other | 8 | 8 | 16
Tumor Type Stratification Factor [Number; unit: Participants]
  Multiple myeloma | 93 | 86 | 179
  Other | 452 | 457 | 909
  Non-small cell lung cancer | 345 | 343 | 688
Previous Skeletal-Related Event Stratification Factor [Number; unit: Participants]
  Yes | 446 | 440 | 886
  No | 444 | 446 | 890
Systematic Anti-Cancer Therapy Stratification Factor [Number; unit: Participants]
  Yes | 747 | 746 | 1493
  No | 143 | 140 | 283

OUTCOME MEASURES:

1. Primary Outcome: Time to the First On-Study Skeletal-Related Event (Non-Inferiority)
Description: Time to the first on-study skeletal-related event (SRE) using a non-inferiority analysis. Median was estimated using the Kaplan-Meier method.
Time Frame: up to 33 months
Population: Full Analysis Set, composed of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 890 | 886
Days | 496.0 [371.00 to 589.00] | 625.0 [456.00 to NA] — Upper limit could not be estimated due to the low number of events
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Non-Inferiority or Equivalence — A synthesis approach was used for a non-inferiority test of the hypothesis that denosumab preserves at least 50% of the effect of zoledronic acid vs. placebo; p = 0.0007, Regression, Cox; Stratified by tumor type, previous skeletal-related event, and systematic anti-cancer therapy; Hazard Ratio (HR) = 0.84, 95% CI [0.71 to 0.98]

2. Secondary Outcome: Time to First On-Study Skeletal-Related Event (Superiority)
Description: Time to first on-study skeletal-related event (SRE) using a test for superiority. Median was estimated using the Kaplan-Meier method.
Time Frame: up to 33 months
Population: Full Analysis Set, composed of all randomized participants.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 890 | 886
Days | 496.0 [371.00 to 589.00] | 625.0 [456.00 to NA] — Upper limit could not be estimated due to the low number of events.
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Superiority or Other; p = 0.060, Regression, Cox; P-value was adjusted for multiplicity according to a hierarchical testing strategy and Hochberg procedure; Hazard Ratio (HR) = 0.84, 95% CI [0.71 to 0.98] — Stratified by tumor type, previous skeletal-related event, and systematic anti-cancer therapy

3. Secondary Outcome: Time to the First-and-Subsequent On-Study Skeletal-Related Event
Description: Time to the first-and-subsequent on-study skeletal-related event (SRE) using multiple event analysis. To be considered a subsequent SRE, the event must occur at least 21 days after the previous SRE.
  This outcome measure utilizes multiple event times, was analyzed based on a proportional mean model, and is therefore more appropriately summarized by the cumulative mean number of events.
Time Frame: up to 33 months
Population: Full Analysis Set, composed of all randomized participants
Measure: Number; unit: Events
Arm/Group | Zoledronic Acid | Denosumab
Number analyzed (Participants) | 890 | 886
Events | 436 | 392
Statistical Analysis 1: Comparison: Zoledronic Acid vs Denosumab; Test type: Superiority or Other; p = 0.145, Anderson-Gill model; P-value was adjusted for multiplicity according to a hierarchical testing strategy and Hochberg procedure; Hazard Ratio (HR) = 0.90, 95% CI [0.77 to 1.04] — Stratified by tumor type, previous skeletal-related event, and systematic anti-cancer therapy

ADVERSE EVENTS:
Time Frame: up to 2 years 9 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Zoledronic Acid 4 mg Q4W | Denosumab 120 mg Q4W
Serious Adverse Events (participants affected / at risk) | 581/878 | 552/878
Other Adverse Events (participants affected / at risk) | 767/878 | 751/878
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4 mg Q4W (N=878) | Denosumab 120 mg Q4W (N=878)
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 49 | 25
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1
Bone marrow failure (Blood and lymphatic system disorders) | 1 | 1
Coagulopathy (Blood and lymphatic system disorders) | 2 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 | 0
Erythropenia (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 31 | 21
Granulocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hyperviscosity syndrome (Blood and lymphatic system disorders) | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 6 | 3
Neutropenia (Blood and lymphatic system disorders) | 11 | 14
Pancytopenia (Blood and lymphatic system disorders) | 11 | 7
Retroperitoneal lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 23 | 17
Acute coronary syndrome (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 3 | 3
Angina pectoris (Cardiac disorders) | 0 | 3
Angina unstable (Cardiac disorders) | 0 | 1
Arrhythmia (Cardiac disorders) | 0 | 4
Arrhythmia supraventricular (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 7 | 7
Atrial flutter (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac arrest (Cardiac disorders) | 3 | 12
Cardiac disorder (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 5 | 10
Cardiac failure acute (Cardiac disorders) | 1 | 2
Cardiac failure congestive (Cardiac disorders) | 3 | 4
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 3 | 4
Cardio-respiratory distress (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Cardiopulmonary failure (Cardiac disorders) | 9 | 8
Congestive cardiomyopathy (Cardiac disorders) | 0 | 1
Extrasystoles (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 0 | 1
Left ventricular failure (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 4 | 3
Myocardial ischaemia (Cardiac disorders) | 2 | 1
Palpitations (Cardiac disorders) | 1 | 0
Paroxysmal arrhythmia (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 5 | 6
Pericarditis (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 2 | 3
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 1
Goitre (Endocrine disorders) | 1 | 0
Hypopituitarism (Endocrine disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Diplopia (Eye disorders) | 1 | 1
Retinal vein occlusion (Eye disorders) | 0 | 1
Vision blurred (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 17 | 18
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 5
Aphagia (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 6 | 4
Caecitis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 1
Colonic polyp (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 9 | 4
Diarrhoea (Gastrointestinal disorders) | 13 | 14
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Dysphagia (Gastrointestinal disorders) | 5 | 7
Enteritis (Gastrointestinal disorders) | 1 | 0
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 1 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1
Faecal incontinence (Gastrointestinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 2 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 8 | 3
Gastrointestinal hypomotility (Gastrointestinal disorders) | 2 | 0
Haematemesis (Gastrointestinal disorders) | 2 | 4
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 4 | 4
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 8
Intestinal perforation (Gastrointestinal disorders) | 2 | 2
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Mechanical ileus (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 16 | 14
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 2
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 2 | 1
Pneumoperitoneum (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 2
Retching (Gastrointestinal disorders) | 0 | 1
Sigmoiditis (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 1
Subileus (Gastrointestinal disorders) | 0 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 24 | 21
Adverse event (General disorders) | 1 | 0
Asthenia (General disorders) | 16 | 21
Catheter related complication (General disorders) | 1 | 0
Chest discomfort (General disorders) | 2 | 1
Chest pain (General disorders) | 10 | 14
Chills (General disorders) | 1 | 0
Death (General disorders) | 8 | 6
Disease progression (General disorders) | 13 | 8
Euthanasia (General disorders) | 0 | 1
Fatigue (General disorders) | 6 | 11
Feeling abnormal (General disorders) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 38 | 26
Generalised oedema (General disorders) | 0 | 1
Hernia (General disorders) | 1 | 0
Hyperpyrexia (General disorders) | 0 | 1
Inflammation of wound (General disorders) | 0 | 1
Local swelling (General disorders) | 0 | 2
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 2 | 2
Multi-organ failure (General disorders) | 8 | 10
Oedema (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 7 | 5
Organ failure (General disorders) | 2 | 1
Pain (General disorders) | 6 | 12
Performance status decreased (General disorders) | 8 | 3
Pyrexia (General disorders) | 21 | 26
Sudden death (General disorders) | 0 | 1
Suprapubic pain (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 2 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 4 | 2
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 1
Hepatorenal failure (Hepatobiliary disorders) | 1 | 2
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 2
Jaundice (Hepatobiliary disorders) | 1 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Liver disorder (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 3
Hypersensitivity (Immune system disorders) | 0 | 1
Abdominal infection (Infections and infestations) | 0 | 1
Abdominal wall infection (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1
Arthritis bacterial (Infections and infestations) | 1 | 0
Aspergillosis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Bacterial infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 0 | 1
Brain abscess (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 3 | 3
Bronchopneumonia (Infections and infestations) | 4 | 2
Catheter related infection (Infections and infestations) | 1 | 0
Cavernous sinus thrombosis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 5 | 5
Clostridial infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 1
Empyema (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 1 | 0
Fungal skin infection (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastritis fungal (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 5 | 5
Gastrointestinal infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 2 | 2
Influenza (Infections and infestations) | 1 | 0
Kidney infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 5 | 5
Localised infection (Infections and infestations) | 1 | 2
Lower respiratory tract infection (Infections and infestations) | 4 | 0
Lung abscess (Infections and infestations) | 2 | 2
Lung infection (Infections and infestations) | 1 | 6
Mastoiditis (Infections and infestations) | 0 | 2
Nasopharyngitis (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 2
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Osteomyelitis acute (Infections and infestations) | 0 | 1
Parotitis (Infections and infestations) | 0 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 1 | 1
Pneumonia (Infections and infestations) | 44 | 52
Pneumonia haemophilus (Infections and infestations) | 1 | 0
Pneumonia klebsiella (Infections and infestations) | 2 | 0
Pneumonia staphylococcal (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pulmonary mycosis (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1
Purulent discharge (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 0 | 1
Rectal abscess (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 8 | 4
Salmonellosis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 11 | 16
Septic shock (Infections and infestations) | 4 | 6
Sinusitis (Infections and infestations) | 1 | 2
Skin infection (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 9 | 9
Urinary tract infection bacterial (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 3 | 2
Viral infection (Infections and infestations) | 0 | 1
Viral pharyngitis (Infections and infestations) | 0 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1
Collapse of lung (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Device dislocation (Injury, poisoning and procedural complications) | 0 | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 1
Femur fracture (Injury, poisoning and procedural complications) | 7 | 5
Fractured ischium (Injury, poisoning and procedural complications) | 1 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 3 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Ilium fracture (Injury, poisoning and procedural complications) | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Lung injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural discharge (Injury, poisoning and procedural complications) | 0 | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1 | 0
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Stent-graft endoleak (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 2 | 4
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 1
Traumatic brain injury (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood calcium decreased (Investigations) | 1 | 0
Blood creatinine abnormal (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 3 | 4
Blood potassium (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0
Creatinine renal clearance decreased (Investigations) | 0 | 1
Haemoglobin decreased (Investigations) | 3 | 0
Monoclonal immunoglobulin present (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Platelet count increased (Investigations) | 0 | 1
Sputum abnormal (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 1
White blood cell count decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 7 | 6
Cachexia (Metabolism and nutrition disorders) | 10 | 4
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 34 | 35
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 2 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 8 | 12
Hypoglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 6 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 2
Marasmus (Metabolism and nutrition disorders) | 1 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 19 | 15
Bone pain (Musculoskeletal and connective tissue disorders) | 15 | 11
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint crepitation (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 5
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bile duct cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Cervix cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 6
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 100 | 103
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to abdominal cavity (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 | 9
Metastases to bone marrow (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 44 | 43
Metastases to gastrointestinal tract (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 13 | 16
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Metastases to rectum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 7
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic carcinoma of the bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Paraneoplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pharyngeal neoplasm benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1
Amnesia (Nervous system disorders) | 0 | 1
Apraxia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Cerebral artery embolism (Nervous system disorders) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 4 | 2
Cerebrovascular accident (Nervous system disorders) | 2 | 5
Cervical cord compression (Nervous system disorders) | 1 | 1
Cervical root pain (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 7 | 5
Coma uraemic (Nervous system disorders) | 0 | 1
Convulsion (Nervous system disorders) | 5 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Diplegia (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 3 | 4
Dysarthria (Nervous system disorders) | 1 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Epiduritis (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 3 | 2
Facial palsy (Nervous system disorders) | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 3
Hemiparesis (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 1 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 2 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 2
Lethargy (Nervous system disorders) | 3 | 0
Loss of consciousness (Nervous system disorders) | 3 | 1
Mental impairment (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 0
Monoplegia (Nervous system disorders) | 1 | 1
Motor dysfunction (Nervous system disorders) | 1 | 0
Nerve root compression (Nervous system disorders) | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1
Neuritis (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 1 | 1
Neurotoxicity (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 3
Paraparesis (Nervous system disorders) | 5 | 5
Paraplegia (Nervous system disorders) | 3 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 2 | 3
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy (Nervous system disorders) | 0 | 1
Polyneuropathy alcoholic (Nervous system disorders) | 0 | 1
Psychomotor skills impaired (Nervous system disorders) | 0 | 1
Sensory disturbance (Nervous system disorders) | 0 | 1
Sensory loss (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 1 | 2
Speech disorder (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 26 | 27
Syncope (Nervous system disorders) | 8 | 3
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 2 | 3
Completed suicide (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 9 | 4
Emotional distress (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 9 | 4
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 | 1
Anuria (Renal and urinary disorders) | 2 | 2
Azotaemia (Renal and urinary disorders) | 0 | 1
Bladder mass (Renal and urinary disorders) | 1 | 0
Bladder obstruction (Renal and urinary disorders) | 0 | 1
Bladder pain (Renal and urinary disorders) | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 2 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 2 | 8
Hydronephrosis (Renal and urinary disorders) | 2 | 1
Nephroangiosclerosis (Renal and urinary disorders) | 1 | 0
Oliguria (Renal and urinary disorders) | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 13 | 10
Renal failure acute (Renal and urinary disorders) | 15 | 10
Renal impairment (Renal and urinary disorders) | 2 | 0
Urethral obstruction (Renal and urinary disorders) | 1 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 2 | 0
Urinary retention (Renal and urinary disorders) | 9 | 3
Urinary tract disorder (Renal and urinary disorders) | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
Orchitis noninfective (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 2 | 4
Uterine haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 54 | 55
Dyspnoea at rest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 9 | 11
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 7
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 27 | 23
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 18 | 19
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 40 | 45
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Lichenoid keratosis (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Immobile (Social circumstances) | 1 | 0
Abdominal wall operation (Surgical and medical procedures) | 1 | 0
Medical device removal (Surgical and medical procedures) | 1 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 1
Aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm (Vascular disorders) | 1 | 0
Aortic occlusion (Vascular disorders) | 1 | 0
Arterial thrombosis (Vascular disorders) | 1 | 0
Arteritis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 13 | 15
Embolism (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 1 | 1
Haemorrhage (Vascular disorders) | 2 | 2
Hypertension (Vascular disorders) | 2 | 1
Hypertensive crisis (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 6 | 9
Hypovolaemic shock (Vascular disorders) | 2 | 1
Jugular vein thrombosis (Vascular disorders) | 2 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 2 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1
Peripheral artery aneurysm (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 0 | 1
Subclavian vein thrombosis (Vascular disorders) | 1 | 1
Superior vena caval occlusion (Vascular disorders) | 2 | 2
Thrombosis (Vascular disorders) | 3 | 1
Vena cava thrombosis (Vascular disorders) | 2 | 0
Venous thrombosis (Vascular disorders) | 1 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Zoledronic Acid 4 mg Q4W (N=878) | Denosumab 120 mg Q4W (N=878)
Anaemia (Blood and lymphatic system disorders) | 264 | 234
Leukopenia (Blood and lymphatic system disorders) | 68 | 50
Neutropenia (Blood and lymphatic system disorders) | 100 | 90
Thrombocytopenia (Blood and lymphatic system disorders) | 86 | 90
Abdominal pain (Gastrointestinal disorders) | 86 | 84
Abdominal pain upper (Gastrointestinal disorders) | 38 | 47
Constipation (Gastrointestinal disorders) | 209 | 188
Diarrhoea (Gastrointestinal disorders) | 165 | 163
Nausea (Gastrointestinal disorders) | 260 | 244
Vomiting (Gastrointestinal disorders) | 167 | 174
Asthenia (General disorders) | 171 | 156
Chest pain (General disorders) | 85 | 92
Fatigue (General disorders) | 216 | 203
Mucosal inflammation (General disorders) | 47 | 43
Oedema peripheral (General disorders) | 135 | 106
Pain (General disorders) | 47 | 47
Pyrexia (General disorders) | 170 | 125
Urinary tract infection (Infections and infestations) | 44 | 38
Rib fracture (Injury, poisoning and procedural complications) | 46 | 39
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 44 | 35
Weight decreased (Investigations) | 105 | 99
Anorexia (Metabolism and nutrition disorders) | 190 | 163
Dehydration (Metabolism and nutrition disorders) | 45 | 42
Hypocalcaemia (Metabolism and nutrition disorders) | 47 | 88
Hypokalaemia (Metabolism and nutrition disorders) | 63 | 53
Arthralgia (Musculoskeletal and connective tissue disorders) | 137 | 124
Back pain (Musculoskeletal and connective tissue disorders) | 183 | 169
Bone pain (Musculoskeletal and connective tissue disorders) | 149 | 137
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 49 | 53
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 95 | 92
Pain in extremity (Musculoskeletal and connective tissue disorders) | 128 | 121
Dizziness (Nervous system disorders) | 72 | 67
Headache (Nervous system disorders) | 93 | 99
Neuropathy peripheral (Nervous system disorders) | 42 | 46
Paraesthesia (Nervous system disorders) | 59 | 45
Anxiety (Psychiatric disorders) | 56 | 73
Depression (Psychiatric disorders) | 56 | 62
Insomnia (Psychiatric disorders) | 93 | 89
Cough (Respiratory, thoracic and mediastinal disorders) | 151 | 172
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 171 | 193
Alopecia (Skin and subcutaneous tissue disorders) | 62 | 48
Rash (Skin and subcutaneous tissue disorders) | 75 | 67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.